CLINICAL TRIAL: NCT04725552
Title: Testing the Feasibility of Pragmatic Case Finding and a Supplemental Digital Intervention for Alcohol-related Health Problems in General Practice
Brief Title: Identifying and Managing Alcohol-related Health Problems in General Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: University of Oslo (Other); Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 8/2020
Record Dates: First submitted 2020-07-27; First posted 2021-01-26 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-09

CONDITIONS: Alcohol-Related Disorders; Alcohol Problem; Alcohol Drug Interaction; Alcohol Use Disorder
Keywords: General practice; Feasibility; Implementation
MeSH Terms: conditions — Alcohol-Related Disorders; Alcoholism

STUDY DESIGN:
Intervention Model Description: Feasibility study of a digital intervention supporting change in alcohol consumption for patients in general practice. The digital intervention is a supplement to usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: 'Change' - an e-health intervention — The aim of the e-health intervention is to support the patient's change process and facilitate the doctor's ability to help. We plan for a web-application instead of a native application. A web-application enables use from mobile devices and from computers and is thus not dependent on a specific mode or system. Before including patients (postponed to September 2020 because of the Corona-virus pandemic), about 30 members of the general public have tested the e-health intervention.

SUMMARY:
The overall purpose of the proposed research is to increase patients' and general practitioners' (GPs') awareness of alcohol as a relevant factor for a wide variety of health problems in general practice, and enable earlier help and treatment. To achieve this, the investigators aim to test the feasibility of a pragmatic strategy for identification of alcohol-related health problems, and the feasibility of a web-based intervention between consultations, as a supplement to usual care in general practice.

DETAILED DESCRIPTION:
Alcohol use is a major health problem, and there is a strong need for improved identification of and interventions for alcohol-related health problems. These constitute somatic and neuropsychiatric health problems, caused, precipitated, or complicated by alcohol use.

The investigators will especially recruit patients in late adulthood (60+), as this group may experience more barriers with digital interventions, and will have more health problems potentially affected by alcohol. The investigators have developed the identification strategy and the interventions in close collaboration with key stakeholders: patients and health care professionals.

The aim is to test the feasibility of interventions for hazardous (a quantity or pattern placing patients at risk for adverse health events) and harmful alcohol consumption (consumption resulting in adverse events), with two distinct components, namely pragmatic case finding and a digital self-administered intervention (called Endre) for use between consultations. The study will focus mainly on aspects related to acceptability, demand, implementation and practicality. The results from this feasibility study may give valuable knowledge on how this treatment approach should be adapted and implemented, and will indicate whether a full-scale RCT is warranted. This study is testing the feasibility of interventions intended to facilitate change for both patients (reduced alcohol consumption) and for physicians (improved addressing of alcohol and improved intervention delivery).

ELIGIBILITY:
Inclusion Criteria:

* Registered patient with participating clinic, accepting that alcohol may be relevant for his/her health problem and wanting to participate

Exclusion Criteria:

* None, except age

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The number of patients offered the web-based intervention | Three months from start date
The number of patients completing baseline registration | Six months from start date
The number of patients using the intervention for at least one week | Six months from start date
The number of patients using the intervention for at least four weeks | Six months from start date

SECONDARY OUTCOMES:
Changes alcohol consumption (AUDIT-C) | Three months from completed baseline registration
  Changes in weekly alcohol consumption and binge drinking between baseline and 3 months
Changes in quality of life (RAND12) | Three months from completed baseline registration
  Changes in quality of life between baseline and 3 months
Changes in mental distress (SCL5) | Three months from completed baseline registration
  Changes in mental distress between baseline and 3 months
Changes in sleeping (Bergen Insomnia Scale) | Three months from completed baseline registration
  Changes in sleeping between baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Torgeir G Lid, MD PhD, Principal Investigator — Helse Stavanger HF
Locations (4):
- Norway (4):
  - Sagene Lokalmedisinske senter, Oslo
  - Stavanger Medisinske Senter, Stavanger
  - Nytorget legesenter, Stavanger
  - Hillevågsdoktoren, Stavanger

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Potthoff S, Brendryen H, Bosnic H, Bhardwaj-Gosling R, Iden KR, Nja ALM, O'Donnell A, Lid TG. Implementing pragmatic case finding to address alcohol use in general practice: a mixed methods feasibility study. Scand J Prim Health Care. 2026 Dec;44(1):2598835. doi: 10.1080/02813432.2025.2598835. Epub 2025 Dec 19. PMID 41414920